CLINICAL TRIAL: NCT01102777
Title: Effectiveness of an Automated Walking Program Targeting Veterans With COPD
Brief Title: Stepping up to Health - for Veterans With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 09-366
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: internet; walking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Other): Control group, instructed to wear the pedometer but not provided with walking goals or instruction.
  Interventions: Other: Usual Care
- Internet-mediated Walking Program (Other): participants in the intervention arm are asked to participate in a walking program
  automated internet-mediated walking program: intervention participants are encouraged to walk daily to their step-count goal while wearing a pedometer provided by the study that will measure their daily step-counts. They are also encouraged to log into their personally tailored website to upload their step counts and obtain other information about the study and progress
  Interventions: Behavioral: automated internet-mediated walking program

INTERVENTIONS:
Behavioral: automated internet-mediated walking program — intervention participants are encouraged to walk daily to their step-count goal while wearing a pedometer provided by the study that will measure their daily step-counts. They are also encouraged to log into their personally tailored website to upload their step counts and obtain other information about the study and progress
  Arms: Internet-mediated Walking Program
Other: Usual Care — Control group, instructed to wear the pedometer but not provided with walking goals or instruction.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to assess the efficacy of an internet-mediated pedometer based intervention that is designed to increase walking and improve function among veterans with chronic obstructive pulmonary disease (COPD). The Specific Aims are: 1) to test the effectiveness of an automated internet-mediated walking program for veterans with COPD with a primary outcome of improvement in health-related quality of life at four-months and at one year in a randomized controlled trial (RCT) with a wait list control. 2) to estimate the effect of internet-mediated walking program for veterans with COPD on all cause days of hospitalization over one year following randomization. 3) to compare intervention reach, participation and satisfaction outcomes between rural and urban veterans among those randomized to the intervention arm. The long-term objective of this research is to develop, evaluate and disseminate effective, low-cost interventions that improve quality of life for veterans, particularly rural veterans, managing complex chronic conditions.

DETAILED DESCRIPTION:
Background:

Low levels of physical activity are common in patients with chronic obstructive pulmonary disease (COPD), and a sedentary lifestyle is associated with poor outcomes including increased mortality, frequent hospitalizations, and poor health-related quality of life. Individuals with COPD who undergo a facility-based, exercise-focused pulmonary rehabilitation program experience significant improvements in health related quality of life, dyspnea, and exercise tolerance as well as reduced rates of hospitalization. Unfortunately, only a small percent of individuals with COPD who could benefit from pulmonary rehabilitation have access to and participate in such programs. Moreover, the benefits of short-term pulmonary rehabilitation programs tend to diminish rapidly after the program ends. Rural veterans are less likely to have access to facility-based pulmonary rehabilitation than urban veterans. Health related quality of life in rural veterans with COPD is significantly worse than for veterans with COPD who live in urban areas.

Objectives:

The primary objective of this study was to assess the efficacy of an Internet-mediated, pedometer-based intervention designed to increase walking and health related quality of life for Veterans with COPD. The specific aims of this randomized controlled trial (RCT) with a wait list control were: 1) To test the effectiveness of an automated internet-mediated walking program for veterans with COPD with a primary outcome of improvement in health related quality of life at four months and at one year; 2) to estimate the effect of the internet-mediated walking program for veterans with COPD on all cause days of hospitalization over one year following randomization; and 3) to compare intervention reach, participation and satisfaction outcomes between rural and urban veterans among those randomized to the intervention arm.

Methods:

Participants were followed for 12 months to investigate the efficacy of the intervention in assisting patients with initiating and maintaining a regular walking program and improving health related quality of life. Eligible and consented patients wore a pedometer to obtain one week of baseline data and then were randomized on a 2:1 ratio to Taking Healthy Steps or to a wait list control. The intervention arm received iterative step-count feedback; individualized step-count goals, motivational and informational messages, and access to an online community. Wait list controls were notified that they were enrolled, but that their intervention would start in one year; however, they kept the pedometer and had access to a static webpage. Both groups completed on-line survey assessments at baseline, 4, and 12 months, and were asked to report adverse events on a regular basis. The primary outcome was changes in health related quality of life, as measured using the St George's Respiratory Questionnaire (SGRQ), a disease-specific instrument in patients with COPD. Secondary outcomes included days of hospitalization during the one-year intervention period, changes in average daily steps as measured using the study pedometer, self-reported dyspnea, intervention reach, and adverse event rates. The analysis was conducted based [on the original randomized treatment assignment regardless of participation (an intent-to-treat analysis) and included both a complete case analysis as well as an all case analysis using a linear mixed-effects model. Between-group differences in change scores (4 months or 12 months) were estimated after adjusting for baseline values of the outcome variables.

Status:

This study is completed. Data analysis and manuscript preparation continue.

ELIGIBILITY:
Inclusion Criteria:

* Adult >= 40 years old
* Diagnosis of COPD, emphysema or chronic bronchitis
* Able to walk a minimum of one block
* Sedentary, defined by less than 150 minutes of self-reported physical activity per week
* Have a doctor or primary care provider in the VA who can provide medical clearance
* Competent to give informed consent
* Must be a regular email user (check weekly)
* Have access to a computer with an internet connection, a USB port, and Windows XP or Vista

Exclusion Criteria:

* Diagnosis codes of quadriplegia and paraplegia or pregnancy-related diagnoses or procedures within the previous year will be excluded from potential participant pool

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline R Richardson, MD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Ney JP, Robinson SA, Richardson CR, Moy ML. Can Technology-Based Physical Activity Programs for Chronic Obstructive Pulmonary Disease Be Cost-Effective? Telemed J E Health. 2021 Nov;27(11):1288-1292. doi: 10.1089/tmj.2020.0398. Epub 2021 Feb 24. PMID 33625893
- [Derived] Moy ML, Martinez CH, Kadri R, Roman P, Holleman RG, Kim HM, Nguyen HQ, Cohen MD, Goodrich DE, Giardino ND, Richardson CR. Long-Term Effects of an Internet-Mediated Pedometer-Based Walking Program for Chronic Obstructive Pulmonary Disease: Randomized Controlled Trial. J Med Internet Res. 2016 Aug 8;18(8):e215. doi: 10.2196/jmir.5622. PMID 27502583
- [Derived] Moy ML, Collins RJ, Martinez CH, Kadri R, Roman P, Holleman RG, Kim HM, Nguyen HQ, Cohen MD, Goodrich DE, Giardino ND, Richardson CR. An Internet-Mediated Pedometer-Based Program Improves Health-Related Quality-of-Life Domains and Daily Step Counts in COPD: A Randomized Controlled Trial. Chest. 2015 Jul;148(1):128-137. doi: 10.1378/chest.14-1466. PMID 25811395
- [Derived] Martinez CH, Moy ML, Nguyen HQ, Cohen M, Kadri R, Roman P, Holleman RG, Kim HM, Goodrich DE, Giardino ND, Richardson CR. Taking Healthy Steps: rationale, design and baseline characteristics of a randomized trial of a pedometer-based Internet-mediated walking program in veterans with chronic obstructive pulmonary disease. BMC Pulm Med. 2014 Feb 3;14:12. doi: 10.1186/1471-2466-14-12. PMID 24491137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted entirely through mail, phone, or internet. Recruitment start was December 2011.
Pre-assignment Details: Randomization required Medical Clearance, the completed Baseline Survey, and valid baseline pedometer data. While 307 participants were Consented, only 239 were randomized. The top three reasons for not being randomized were: Pt withdrew prior (23) Failed to submit Medical Clearance and pedometer data (19) or failed to submit Baseline survey (9).
Period: Overall Study
Arm/Group | Usual Care | Internet-mediated Walking Program
Started | 84 | 155
Completed | 75 | 139
Not Completed | 9 | 16
Not completed — Death | 2 | 6
Not completed — Lost to Follow-up | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Internet-mediated Walking Program | Total
Number analyzed (Participants) | 84 | 155 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.2) | 66.9 (8.7) | 66.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 77 | 147 | 224
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 3 | 7 | 10
  White | 79 | 143 | 222
  Other/combined | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 84 | 155 | 239
St George's Respiratory Questionnaire (SGRQ) [Mean (Standard Deviation); unit: units on a scale] — Reflected here is the St George's Respiratory Questionnaire (SGRQ) Total Score. Scores range from 0 to 100, with higher scores indicating more limitations.
  units on a scale | 46.8 (15.6) | 45.5 (15.4) | 46.0 (15.4)
Modified Medical Research Council (MMRC) Dyspnea score [Number; unit: participants] — The Modified Medical Research Council Dyspnea Scale, or MMRC, uses a simple grading system to assess a patient's level of dyspnea -- shortness of breath. Scores range from 0 to 4, with 4 indicating more limitations to daily activities.
  participants
    MMRS Dyspnea Score 0-1 | 57 | 109 | 166
    MMRS Dyspnea Score 2-4 | 27 | 46 | 73
Baseline daily step count; mean [Mean (Standard Deviation); unit: steps] | 3521 (2058) | 3484 (2309) | 3497 (2220)

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Respiratory-Specific Quality of Life
Description: Change in St. George's Respiratory Questionnaire (SGRQ) Total Score from Baseline to four months. (Scores range from 0 to 100, with higher scores indicating more limitations.)
Time Frame: four months from randomization
Population: One Intervention participant was dropped from analysis due to being an extreme outlier. In addition, not all participants had complete SGRQ data at both time points for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Internet-mediated Walking Program
Number analyzed (Participants) | 77 | 144
units on a scale | -0.8 (10.9) | -3.2 (11.1)
Statistical Analysis 1: Comparison: Usual Care vs Internet-mediated Walking Program; Test type: Superiority or Other; p = 0.142, Regression, Linear; Adjusted for baseline value of outcome, MMRC dyspnea score, and urban versus rural residence

2. Primary Outcome: Self-Reported Respiratory-Specific Quality of Life
Description: Change in St. George's Respiratory Questionnaire (SGRQ) Total Score from Baseline to twelve months. (Scores range from 0 to 100, with higher scores indicating more limitations.)
Time Frame: twelve months from randomization
Population: One Intervention participant was dropped from analysis due to being an extreme outlier.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Internet-mediated Walking Program
Number analyzed (Participants) | 84 | 154
units on a scale | -1.4 [-4.1 to 1.3] | -2.5 [-4.5 to -0.6]
Statistical Analysis 1: Comparison: Usual Care vs Internet-mediated Walking Program; Test type: Superiority or Other; p = .502, Mixed Models Analysis; Based on mixed models, adjusting for group, time, group*time interaction, MMRC score, and urban versus rural residence

3. Secondary Outcome: Self Reported Dyspnea
Description: Change in Self Reported Dyspnea from Baseline to 4 months. (Scores range from 0 to 4, with higher scores indicating more shortness of breath. For example, "0 - I only get breathless with strenuous exercise." and "4 - I am too breathless to leave the house or I am breathless when dressing.")
Time Frame: four months from randomization
Population: One Intervention participant was dropped from analysis due to being an extreme outlier. Three Control and ten Intervention were missing values at 4 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Internet-mediated Walking Program
Number analyzed (Participants) | 81 | 144
units on a scale | -.037 (.8) | .035 (.86)
Statistical Analysis 1: Comparison: Usual Care vs Internet-mediated Walking Program; Test type: Superiority or Other; p = .90, Regression, Linear; Adjusted for baseline value and rural residence

4. Secondary Outcome: Self Reported Dyspnea
Description: Change in Self Reported Dyspnea from Baseline to 12 months. (Scores range from 0 to 4, with higher scores indicating more shortness of breath. For example, "0 - I only get breathless with strenuous exercise." and "4 - I am too breathless to leave the house or I am breathless when dressing.")
Time Frame: twelve months from randomization
Population: One Intervention participant was dropped from analysis due to being an extreme outlier. Nine Control and seventeen Intervention participants were missing data at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Internet-mediated Walking Program
Number analyzed (Participants) | 75 | 137
units on a scale | .013 (.88) | .029 (.94)
Statistical Analysis 1: Comparison: Usual Care vs Internet-mediated Walking Program; Test type: Superiority or Other; p = .93, Regression, Linear; Adjusted for baseline value and rural residence

5. Secondary Outcome: Days of Hospitalization
Description: Number of days of all-cause hospitalization during study participation.
Time Frame: during study participation, up to 12 months
Measure: Number; unit: days
Arm/Group | Usual Care | Internet-mediated Walking Program
Number analyzed (Participants) | 84 | 155
days | 86 | 286
Statistical Analysis 1: Comparison: Usual Care vs Internet-mediated Walking Program; Test type: Superiority or Other; p = .08, Zero inflated Poisson regression; Adjusted for age, gender, oxygen use, and arm

6. Secondary Outcome: Change in Average Daily Step Counts
Description: Change in daily step counts compared to baseline and those captured in the final two weeks of the intervention and the two weeks post intervention.
Time Frame: baseline and final two weeks of the intervention and the two weeks post intervention.
Population: One Intervention participant was dropped from analysis due to being an extreme outlier.
Measure: Mean (95% Confidence Interval); unit: steps
Arm/Group | Usual Care | Internet-mediated Walking Program
Number analyzed (Participants) | 84 | 154
steps | 163 [-336 to 661] | 270 [-86 to 626]
Statistical Analysis 1: Comparison: Usual Care vs Internet-mediated Walking Program; Test type: Superiority or Other; p = 0.731, Mixed Models Analysis; Based on mixed models, adjusting for group, time, group*time interaction, MMRC score, and urban versus rural residence

7. Secondary Outcome: Goal Commitment for Intervention Participants
Description: Change in goal commitment for intervention participations on a Likert scale from 1-5, with 1 as "Strongly Disagree" and 5 is "Strongly Agree" to the question, "I am strongly committed to pursuing my step count goal." A negative change value indicates lower goal commitment.
Time Frame: change from four months and twelve months from enrollment
Population: This measure was only assessed on the Intervention group, and only 146 participants answered the question at either time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Internet-mediated Walking Program
Number analyzed (Participants) | 0 | 146
units on a scale |  | -.08 [-.32 to .16]
Statistical Analysis 1: Comparison: Internet-mediated Walking Program; Test type: Superiority or Other; p = .52, Mixed Models Analysis; Based on mixed models, adjusting for time, MMRC score, and urban versus rural residence

8. Secondary Outcome: Study Reach Among Rural Participants
Description: Calculated by dividing the total number of eligible rural responders by the total number of rural responders to create an eligibility rate, then multiplying the eligibility rate with the total number of letters sent to rural individuals to create a possible rural eligible pool. The total number of eligible rural responders was divided by the possible rural eligible pool.
Time Frame: At baseline
Population: number of rural participants.
Measure: Number; unit: percentage of possible eligible rural
Groups:
- Intervention: participants in the intervention arm are asked to participate in a walking program
  automated internet-mediated walking program: intervention participants are encouraged to walk daily to their step-count goal while wearing a pedometer provided by the study that will measure their daily step-counts. They are also encouraged to log into their personally tailored website to upload their step counts and obtain other information about the study and progress
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 37 | 71
percentage of possible eligible rural | 2.5 | 2.5
Statistical Analysis 1: Comparison: Usual Care vs Intervention; The determination of arm occurred after recruitment, and Study Reach is a recruitment value; Test type: Superiority or Other; Mean Difference (Net) = 0

9. Secondary Outcome: Participant Retention
Description: The last valid day of pedometer data or the last login day to the study website for both arms, whichever day was last, from 1-366.
Time Frame: during study participation, up to twelve months
Measure: Mean (95% Confidence Interval); unit: day
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 84 | 154
day | 308.8 [287.9 to 329.6] | 329.6 [314.2 to 345]
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority or Other; p = .11, Regression, Linear; Adjusting for time, MMRC score, and urban versus rural residence

10. Secondary Outcome: Change in Participant Satisfaction
Description: Change in participation satisfaction with the Intervention group from four to twelve months on a Likert scale of 1-5, where 1 is "Definitely True" 5 is "Definitely False" to the question, "I would recommend the Taking Healthy Steps walking program to another person with COPD". A negative change value indicates higher satisfaction score.
Time Frame: four to twelve months of study participation
Population: This was only assessed on Intervention group participants who answered the question at either four or twelve months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 0 | 146
units on a scale |  | -.14 [-.26 to -.03]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority or Other; p = .01, Mixed Models Analysis; Based on mixed models, adjusting for time, MMRC score, and urban versus rural residence

ADVERSE EVENTS:
Time Frame: During study participation, up to twelve months.
Description: Participants could report adverse events at any time. Participants in both groups were also prompted monthly to report new or worsening medical symptoms or problems, whether or not study related. Additionally, data for hospitalizations was gathered from VA medical record
Arm/Group | Usual Care | Internet-mediated Walking Program
Serious Adverse Events (participants affected / at risk) | 19/84 | 44/155
Other Adverse Events (participants affected / at risk) | 39/84 | 90/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=84) | Internet-mediated Walking Program (N=155)
General disorders (General disorders) | 19 (28) | 44 (64) — Serious adverse events during the study period ranged from hospitalizations for planned surgeries to death. All were reviewed and none were found to be study-related. They were reported but not categorized by system.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=84) | Internet-mediated Walking Program (N=155)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (9) | 43 (70)
Cardiac disorders (Cardiac disorders) | 1 (1) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 27 (35) | 39 (156)
Other (General disorders) | 3 (3) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No